CLINICAL TRIAL: NCT00958802
Title: Tissue Engineering Microtia Auricular Reconstruction: in Vitro and in Vivo Studies
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Chia-Che Wu, MD, Taipei medical university- Wan Fang Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 98-WF-PHD-05
Record Dates: First submitted 2009-08-12; First posted 2009-08-13 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: Microtia
Keywords: tissue engineering
MeSH Terms: conditions — Congenital Microtia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Placebo Comparator): Chondrocyte culture with FBS medium
  Interventions: Other: Chondrocyte culture with FBS medium
- Arm B (Experimental): Chondrocyte culture with PRP
  Interventions: Other: Platelet-rich plasma (PRP)

INTERVENTIONS:
Other: Platelet-rich plasma (PRP) — PRP was extracted from total blood and TGF-b1 was used as indicator
  Arms: Arm B
Other: Chondrocyte culture with FBS medium — Microtia chondrocyte culture with FBS medium only
  Arms: Arm A

SUMMARY:
Platelet-rich plasma (PRP) has mixed growth factors such as TGF-ß1 and TGF-ß2, vascular epithelial growth factor (VEGF), platelet-derived growth factor (PDGF), and insulin-like growth factor (IGF). These growth factors appear to play an important role in wound healing and are assumed as promoters of tissue regeneration. Moreover, PRP was used as injectable scaffold seeded with chondrocytes to regenerate cartilage. In their previous study, the investigators concluded that growth factors in PRP can effectively react as a growth factor cocktail to induce human nucleus pulposus proliferation and differentiation, and also promote tissue-engineered nucleus pulposus formation. The investigators also have a hypothesis that PRP can promote tissue-engineered microtia auricular cartilage formation. TGF- ß1 exists in the highest concentration and is more important among all of the growth factors released from PRP. So TGF- ß1 can be used as the core ingredient and the indicator for applying PRP in these studies. The aim of this study was to compare the histological and biochemical character of microtia chondrocytes treated with and without PRP.

ELIGIBILITY:
Inclusion Criteria:

* microtia patient

Exclusion Criteria:

* non microtia patient

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2009-05; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
The aim of this study was to compare the histological and biochemical character of microtia chondrocytes treated with and without PRP. | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Che Wu, MD, Study Chair — Chia-Che Wu
Locations (1):
- Taipei Medical University, Wan Fang Hospital, Taipei, Taiwan